CLINICAL TRIAL: NCT01659554
Title: A Phase II Combined Modality Protocol of Debulking Surgery With Heated Intraoperative Chemotherapy (HIPEC) Followed by Intraperitoneal Chemotherapy for the Treatment of Recurrent Ovarian, Primary Peritoneal and Fallopian Tube Cancers
Brief Title: A Phase II Combined Modality Protocol of Debulking Surgery With HIPEC Followed by Intraperitoneal Chemotherapy for the Treatment of Recurrent Ovarian, Primary Peritoneal & Fallopian Tube Cancers
Acronym: HIPEC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator left institution
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAI1246
Record Dates: First submitted 2012-07-10; First posted 2012-08-08 (Estimated); Results first posted 2015-03-03 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Recurrent Ovarian Cancer; Fallopian Tube Cancer
Keywords: Primary peritoneal
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Cisplatin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Out-Patient Intraperitoneal Chemotherapy (Experimental): Intraoperative (hyperthermic) cisplatin followed by 4 courses of intraperitoneal cisplatin and doxorubicin given on days 1 & 8 during a 3 week cycle.
  Interventions: Drug: Cisplatin; Drug: Doxorubicin

INTERVENTIONS:
Drug: Cisplatin — Cisplatin (75 mg/m2) prepared in 2L normal saline.
  Other Names: cis-diamminedichloroplatinum(II) (CDDP); Platinol; Platinol-AQ
Drug: Doxorubicin — Doxorubicin (25 mg flat dose) prepared in 500 ml dialysis fluid (glucose or icodextrin-based).
  Other Names: hydroxyldaunorubicin; Adriamycin

SUMMARY:
The primary objective of this study is to investigate the feasibility, tolerability and safety of surgical debulking and resection with heated intraoperative chemotherapy (HIPEC) followed by repeated intraperitoneal chemotherapy for treatment of recurrent ovarian, primary peritoneal, and fallopian tube carcinomas.

DETAILED DESCRIPTION:
This is a phase II , open label, single center study of surgery followed by heated intraoperative cisplatin in patients with recurrent ovarian, primary peritoneal or fallopian tube cancers. Approximately twenty patients will receive surgery and intraoperative (hyperthermic) cisplatin followed by four consecutive courses of outpatient intraperitoneal cisplatin and doxorubicin given on days 1 and 8 during a 3 week cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed ovarian, primary peritoneal or fallopian tube carcinoma.
2. Patients must have measurable evidence of recurrent intraabdominal disease based on Computed tomography (CT scan) findings.
3. Patients must fulfill the following with regard to prior chemotherapy:

   1. 4 weeks or greater since conclusion of prior chemotherapy;
   2. Prior intraperitoneal chemotherapy with cisplatin is acceptable; and,
   3. Prior systemic chemotherapy is acceptable.
4. Patients must have a Karnofsky Performance Status of > 70%
5. Patients must have an estimated life expectancy of at least 16 weeks.
6. Patient assurance of study compliance and geographic proximity that allows for adequate follow-up.
7. Patients must have adequate organ function at the screening visit as defined by the following laboratory values:

   Absolute neutrophil count (ANC) ≥1.5 x 109/L Platelet count ≥100 x 109/L Hemoglobin ≥8 g/dL Albumin ≥ 2 g/dL Total Bilirubin ≤ 2.5 x ULN* Alkaline phosphatase ≤ 3.0 x ULN* Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 x ULN Creatinine ≤ 1.5 x ULN
8. Patient must have signed informed consent
9. Patient must be at least 18 years of age
10. Following cytoreductive surgery, patient's residual disease should be no larger than 1cm to Receive HIPEC and continue with normothermic IP chemotherapy

Exclusion criteria:

1. Have active peripheral neuropathy of Grade 2 or greater intensity, as defined by the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE; Version 4).
2. Have experienced myocardial infarction within 6 months prior to enrollment or have New York Hospital Association (NYHA) Class III or IV heart failure (see section 16.4), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
3. Prior radiation therapy within 4 weeks of enrollment.
4. Have uncontrolled active systemic infection requiring therapy.
5. Have a history of allergic reaction attributable to compounds containing boron or mannitol or hypersensitivity reactions to drugs formulated with polysorbate 80.
6. Have had a serious concomitant systemic disorders (including oncologic emergencies) incompatible with the study (at the discretion of the investigator).
7. Have had a "currently active" second malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix are not to be registered. Patients who are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse.
8. Have had any investigational agent within 4 weeks before enrollment into the study.
9. Have a history of a serious medical or psychiatric illness preventing informed consent or, in the opinion of the investigator, would make the patient a poor study candidate.
10. Evidence of extraabdominal metastasis on preinclusion thoracic computed tomography (CT) scans (i.e. brain or chest disease).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharyn Lewin, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled during 10/23/2012 to 08/20/2013.
Groups:
- Intraoperative Cisplatin Followed by IP Chemotherapy: Intraoperative (hyperthermic) cisplatin followed by 4 courses of intraperitoneal cisplatin and doxorubicin given on days 1 & 8 during a 3 week cycle
  Intraoperative (hyperthermic) cisplatin followed by IP Cisplatin; Doxorubicin: Cisplatin 75 mg/m2 at 40.5-42.5 Celsius intraoperatively administered; IP Cisplatin 75 mg/m2 (Day 1) week 1 followed by IP Doxorubicin 25 mg week 2 (day 8) for four sequential 3 week cycles;
Period: Overall Study
Arm/Group | Intraoperative Cisplatin Followed by IP Chemotherapy
Started | 4 (4 subjects enrolled; 4 subjects treated and 4 did not complete protocol schema)
Completed | 0
Not Completed | 4
Not completed — Study Termination | 4

BASELINE CHARACTERISTICS:
Arm/Group | Intraoperative Cisplatin Followed by IP Chemotherapy
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Adverse Event Rate and/or Laboratory Changes
Description: The adverse event rate and laboratory changes will be used to investigate the safety of surgical debulking with heated intraperitoneal chemotherapy (HIPEC) combined with repeated intraperitoneal chemotherapy.
Time Frame: 5 years
Population: zero participants analyzed due to early termination of study
Arm/Group | Intraoperative Cisplatin Followed by IP Chemotherapy
Number analyzed (Participants) | 0

2. Primary Outcome: Toxicity Rating Based on NCI Common Toxicity Criteria
Description: Patients will be rated for toxicity prior to each cycle using the NCI Common Toxicity Criteria (NCICTC; see the CTCAE, Version 4.0).
Time Frame: Up to 5 years
Population: zero participants analyzed due to early termination of study
Arm/Group | Intraoperative Cisplatin Followed by IP Chemotherapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Serum Ca-125 Nadir and/or CT Response (RECIST Criteria)
Description: Efficacy of surgical resection with HIPEC combined with repeated intraperitoneal chemotherapy: The end point will be the objective response rate and progression-free survival as well as the overall survival, if feasible. We will analyze the time to serum Ca 125 nadir and/or CT response based on Recist criteria.
Time Frame: Up to 5 years (survival)
Population: zero participants analyzed due to early termination of study
Arm/Group | Intraoperative Cisplatin Followed by IP Chemotherapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Kaplan-Meier Curves for Patient Overall Survival
Description: Kaplan-Meier analysis will be done using PROC LIFETEST in Statistical Application Software (SAS).
Time Frame: Up to 5 years, survival
Population: zero participants analyzed due to early termination of study
Arm/Group | Intraoperative Cisplatin Followed by IP Chemotherapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Intraoperative Cisplatin Followed by IP Chemotherapy
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intraoperative Cisplatin Followed by IP Chemotherapy (N=4)
Ileus, Grade 3 (Gastrointestinal disorders) | 1 (1)
Grade 2 Abdominal Pain (Infections and infestations) | 1 (1) — due to malfunctional intraperitoneal port
IP drain infection, grade 3 (Infections and infestations) | 1 (1)
Nausea & vomiting (Gastrointestinal disorders) | 1 (1)
No Oliguric Acute Renal Injury (Renal and urinary disorders) | 1 (1)
Urinary Trasct Infection Grade 3 (Renal and urinary disorders) | 1 (1)
Right Shoulder cellulitis (Infections and infestations) | 1 (1)
Fever with catheter related infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Zero participants analyzed due to early termination of study. Adverse Events could not be collected over the pre-specified Time Frame ("5 years") due to study termination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No